CLINICAL TRIAL: NCT03026465
Title: Vessel Injury in Relation With Strut Thickness Assessed by OCT (VISTA): A Comparison of Vascular Injury Induced by a Polymer Free Sirolimus and Probucol Eluting Stent and a Biodegradable-polymer Biolimus-eluting Stent
Brief Title: Vessel Injury in Relation With Strut Thickness Assessed by OCT
Acronym: VISTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Investigacion Interhospitalaria Cardiovascular (Other)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Principal Investigator, Nieves Gonzalo, MD, PhD, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VISTA
Record Dates: First submitted 2016-10-28; First posted 2017-01-20 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coroflex ISAR stent (Experimental): PCI with a polymer-free dual-drug sirolimus- and probucol-eluting stent (Coroflex ISAR stent) with very thin struts (50 µm). During the PCI, an OCT assessment (baseline and post-implantation) will be performed.
  Interventions: Device: Polymer-free stent
- Biomatrix stent (Active Comparator): PCI with a biodegradable-polymer biolimus-eluting stent (Biomatrix stent) with 120 µm struts. During the PCI, an OCT assessment (baseline and post-implantation) will be performed.
  Interventions: Device: Biodegradable-polymer stent

INTERVENTIONS:
Device: Polymer-free stent — PCI using a polymer-free dual-drug sirolimus- and probucol-eluting stent (Coroflex ISAR)
  Other Names: Coroflex ISAR
  Arms: Coroflex ISAR stent
Device: Biodegradable-polymer stent — PCI using a biodegradable-polymer biolimus-eluting stent (Biomatrix)
  Other Names: Biomatrix
  Arms: Biomatrix stent

SUMMARY:
The objective of the present study is to determine the relation between vascular injury induced by the stent and strut thickness.

DETAILED DESCRIPTION:
Thinner struts produce less arterial injury after stent implantation.The objective of the present study is to determine the relation between vascular injury induced by the stent and strut thickness. Vessel injury after stent implantation will be evaluated with optical coherence tomography (OCT). Two stents platforms with different strut thickness (Coroflex ISAR 50 microns and Biomatrix 120 microns) will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Ischemic symptoms or evidence of myocardial ischemia (inducible or spontaneous) in the presence of >50% de novo stenosis located in native coronary vessels

Exclusion Criteria:

* Target lesion located in the left main stem
* STEMI
* Restenosis
* Cardiogenic shock
* Malignancies or other comorbid conditions with life expectancy less than 12 months or that may result in protocol noncompliance
* Known allergy to the study medications (probucol, sirolimus, zotarolimus)
* Pregnancy (present, suspected, or planned)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
OCT-based intimal injury score | Up to 1 day (evaluated after stent implantation)
  OCT-based intimal injury score estimated after implantation of the Coroflex-ISAR and Biomatrix DES

SECONDARY OUTCOMES:
Tissue prolapse area | Up to 1 day (evaluated after stent implantation)
  Tissue prolapse area assessed by OCT after implantation of Coroflex-ISAR and Biomatrix will be measured
Incidence of stent malapposition | Up to 1 day (evaluated after stent implantation)
  Stent apposition after implantation of Coroflex-ISAR and Biomatrix as assessed by OCT
Incidence of stent underexpansion | Up to 1 day (evaluated after stent implantation)
  Stent expansion will be measured with OCT after implantation of Coroflex-ISAR and Biomatrix
Stent symmetry after implantation | Up to 1 day (evaluated after stent implantation)
  Stent symmetry will be measured with OCT after implantation of Coroflex-ISAR and Biomatrix
Baseline plaque type | Up to 1 day (evaluated after stent implantation)
  Baseline plaque type will be assessed by OCT (fibrous, fibrocalcific or lipid-rich)

CONTACTS AND LOCATIONS:
Overall Officials: Nieves Gonzalo, MD, PhD, Study Director — Hospital Clinico San Carlos de Madrid
Locations (3):
- Spain (3):
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sullivan TM, Ainsworth SD, Langan EM, Taylor S, Snyder B, Cull D, Youkey J, Laberge M. Effect of endovascular stent strut geometry on vascular injury, myointimal hyperplasia, and restenosis. J Vasc Surg. 2002 Jul;36(1):143-9. doi: 10.1067/mva.2002.122878. PMID 12096272
- [Background] Hara H, Nakamura M, Palmaz JC, Schwartz RS. Role of stent design and coatings on restenosis and thrombosis. Adv Drug Deliv Rev. 2006 Jun 3;58(3):377-86. doi: 10.1016/j.addr.2006.01.022. Epub 2006 Mar 6. PMID 16650911
- [Background] Farb A, Weber DK, Kolodgie FD, Burke AP, Virmani R. Morphological predictors of restenosis after coronary stenting in humans. Circulation. 2002 Jun 25;105(25):2974-80. doi: 10.1161/01.cir.0000019071.72887.bd. PMID 12081990
- [Background] Rogers C, Edelman ER. Endovascular stent design dictates experimental restenosis and thrombosis. Circulation. 1995 Jun 15;91(12):2995-3001. doi: 10.1161/01.cir.91.12.2995. PMID 7796511
- [Background] Scott NA. Restenosis following implantation of bare metal coronary stents: pathophysiology and pathways involved in the vascular response to injury. Adv Drug Deliv Rev. 2006 Jun 3;58(3):358-76. doi: 10.1016/j.addr.2006.01.015. Epub 2006 Mar 6. PMID 16733073
- [Background] Foin N, Lee RD, Torii R, Guitierrez-Chico JL, Mattesini A, Nijjer S, Sen S, Petraco R, Davies JE, Di Mario C, Joner M, Virmani R, Wong P. Impact of stent strut design in metallic stents and biodegradable scaffolds. Int J Cardiol. 2014 Dec 20;177(3):800-8. doi: 10.1016/j.ijcard.2014.09.143. Epub 2014 Oct 7. PMID 25449502
- [Background] Kolandaivelu K, Swaminathan R, Gibson WJ, Kolachalama VB, Nguyen-Ehrenreich KL, Giddings VL, Coleman L, Wong GK, Edelman ER. Stent thrombogenicity early in high-risk interventional settings is driven by stent design and deployment and protected by polymer-drug coatings. Circulation. 2011 Apr 5;123(13):1400-9. doi: 10.1161/CIRCULATIONAHA.110.003210. Epub 2011 Mar 21. PMID 21422389
- [Background] Foin N, Gutierrez-Chico JL, Nakatani S, Torii R, Bourantas CV, Sen S, Nijjer S, Petraco R, Kousera C, Ghione M, Onuma Y, Garcia-Garcia HM, Francis DP, Wong P, Di Mario C, Davies JE, Serruys PW. Incomplete stent apposition causes high shear flow disturbances and delay in neointimal coverage as a function of strut to wall detachment distance: implications for the management of incomplete stent apposition. Circ Cardiovasc Interv. 2014 Apr;7(2):180-9. doi: 10.1161/CIRCINTERVENTIONS.113.000931. Epub 2014 Mar 18. PMID 24642998
- [Background] Bourantas CV, Papafaklis MI, Kotsia A, Farooq V, Muramatsu T, Gomez-Lara J, Zhang YJ, Iqbal J, Kalatzis FG, Naka KK, Fotiadis DI, Dorange C, Wang J, Rapoza R, Garcia-Garcia HM, Onuma Y, Michalis LK, Serruys PW. Effect of the endothelial shear stress patterns on neointimal proliferation following drug-eluting bioresorbable vascular scaffold implantation: an optical coherence tomography study. JACC Cardiovasc Interv. 2014 Mar;7(3):315-24. doi: 10.1016/j.jcin.2013.05.034. Epub 2014 Feb 13. PMID 24529931
- [Background] Kastrati A, Mehilli J, Dirschinger J, Dotzer F, Schuhlen H, Neumann FJ, Fleckenstein M, Pfafferott C, Seyfarth M, Schomig A. [Intracoronary Stenting and Angiographic Results Strut Thickness Effect on Restenosis Outcome (ISAR-STEREO) Trial]. Vestn Rentgenol Radiol. 2012 Mar-Apr;(2):52-60. Russian. PMID 22730760
- [Background] Pache J, Kastrati A, Mehilli J, Schuhlen H, Dotzer F, Hausleiter J, Fleckenstein M, Neumann FJ, Sattelberger U, Schmitt C, Muller M, Dirschinger J, Schomig A. Intracoronary stenting and angiographic results: strut thickness effect on restenosis outcome (ISAR-STEREO-2) trial. J Am Coll Cardiol. 2003 Apr 16;41(8):1283-8. doi: 10.1016/s0735-1097(03)00119-0. PMID 12706922
- [Background] Joner M, Finn AV, Farb A, Mont EK, Kolodgie FD, Ladich E, Kutys R, Skorija K, Gold HK, Virmani R. Pathology of drug-eluting stents in humans: delayed healing and late thrombotic risk. J Am Coll Cardiol. 2006 Jul 4;48(1):193-202. doi: 10.1016/j.jacc.2006.03.042. Epub 2006 May 5. PMID 16814667
- [Background] Koppara T, Joner M, Bayer G, Steigerwald K, Diener T, Wittchow E. Histopathological comparison of biodegradable polymer and permanent polymer based sirolimus eluting stents in a porcine model of coronary stent implantation. Thromb Haemost. 2012 Jun;107(6):1161-71. doi: 10.1160/TH12-01-0043. Epub 2012 Apr 26. PMID 22535188
- [Background] Finn AV, Joner M, Nakazawa G, Kolodgie F, Newell J, John MC, Gold HK, Virmani R. Pathological correlates of late drug-eluting stent thrombosis: strut coverage as a marker of endothelialization. Circulation. 2007 May 8;115(18):2435-41. doi: 10.1161/CIRCULATIONAHA.107.693739. Epub 2007 Apr 16. PMID 17438147
- [Background] Joner M, Nakazawa G, Finn AV, Quee SC, Coleman L, Acampado E, Wilson PS, Skorija K, Cheng Q, Xu X, Gold HK, Kolodgie FD, Virmani R. Endothelial cell recovery between comparator polymer-based drug-eluting stents. J Am Coll Cardiol. 2008 Jul 29;52(5):333-42. doi: 10.1016/j.jacc.2008.04.030. PMID 18652940
- [Background] Finn AV, Nakazawa G, Joner M, Kolodgie FD, Mont EK, Gold HK, Virmani R. Vascular responses to drug eluting stents: importance of delayed healing. Arterioscler Thromb Vasc Biol. 2007 Jul;27(7):1500-10. doi: 10.1161/ATVBAHA.107.144220. Epub 2007 May 17. PMID 17510464
- [Background] Stefanini GG, Byrne RA, Serruys PW, de Waha A, Meier B, Massberg S, Juni P, Schomig A, Windecker S, Kastrati A. Biodegradable polymer drug-eluting stents reduce the risk of stent thrombosis at 4 years in patients undergoing percutaneous coronary intervention: a pooled analysis of individual patient data from the ISAR-TEST 3, ISAR-TEST 4, and LEADERS randomized trials. Eur Heart J. 2012 May;33(10):1214-22. doi: 10.1093/eurheartj/ehs086. Epub 2012 Mar 24. PMID 22447805
- [Background] Smits PC, Hofma S, Togni M, Vazquez N, Valdes M, Voudris V, Slagboom T, Goy JJ, Vuillomenet A, Serra A, Nouche RT, den Heijer P, van der Ent M. Abluminal biodegradable polymer biolimus-eluting stent versus durable polymer everolimus-eluting stent (COMPARE II): a randomised, controlled, non-inferiority trial. Lancet. 2013 Feb 23;381(9867):651-60. doi: 10.1016/S0140-6736(12)61852-2. Epub 2013 Jan 30. PMID 23374650
- [Background] Vlachojannis GJ, Smits PC, Hofma SH, Togni M, Vazquez N, Valdes M, Voudris V, Puricel S, Slagboom T, Goy JJ, den Heijer P, van der Ent M. Long-term clinical outcomes of biodegradable polymer biolimus-eluting stents versus durable polymer everolimus-eluting stents in patients with coronary artery disease: three-year follow-up of the COMPARE II (Abluminal biodegradable polymer biolimus-eluting stent versus durable polymer everolimus-eluting stent) trial. EuroIntervention. 2015 Jul;11(3):272-9. doi: 10.4244/EIJV11I3A53. PMID 26196753
- [Background] Otsuka F, Cheng Q, Yahagi K, Acampado E, Sheehy A, Yazdani SK, Sakakura K, Euller K, Perkins LEL, Kolodgie FD, Virmani R, Joner M. Acute Thrombogenicity of a Durable Polymer Everolimus-Eluting Stent Relative to Contemporary Drug-Eluting Stents With Biodegradable Polymer Coatings Assessed Ex Vivo in a Swine Shunt Model. JACC Cardiovasc Interv. 2015 Aug 17;8(9):1248-1260. doi: 10.1016/j.jcin.2015.03.029. PMID 26292590
- [Background] Otsuka F, Yahagi K, Ladich E, Kutys R, Alexander R, Fowler D, Virmani R, Joner M. Hypersensitivity reaction in the US Food and Drug Administration-approved second-generation drug-eluting stents: histopathological assessment with ex vivo optical coherence tomography. Circulation. 2015 Jan 20;131(3):322-4. doi: 10.1161/CIRCULATIONAHA.114.012658. No abstract available. PMID 25601953
- [Background] Massberg S, Byrne RA, Kastrati A, Schulz S, Pache J, Hausleiter J, Ibrahim T, Fusaro M, Ott I, Schomig A, Laugwitz KL, Mehilli J; Intracoronary Stenting and Angiographic Results: Test Efficacy of Sirolimus- and Probucol-Eluting Versus Zotarolimus- Eluting Stents (ISAR-TEST 5) Investigators. Polymer-free sirolimus- and probucol-eluting versus new generation zotarolimus-eluting stents in coronary artery disease: the Intracoronary Stenting and Angiographic Results: Test Efficacy of Sirolimus- and Probucol-Eluting versus Zotarolimus-eluting Stents (ISAR-TEST 5) trial. Circulation. 2011 Aug 2;124(5):624-32. doi: 10.1161/CIRCULATIONAHA.111.026732. Epub 2011 Jul 18. PMID 21768546
- [Background] Alfonso F, Sandoval J, Perez-Vizcayno MJ, Cardenas A, Gonzalo N, Jimenez-Quevedo P, Ibanez B, Nunez-Gil I, Rivero F, Escaned J, Fernandez-Ortiz A, Macaya C. Mechanisms of balloon angioplasty and repeat stenting in patients with drug-eluting in-stent restenosis. Int J Cardiol. 2015 Jan 15;178:213-20. doi: 10.1016/j.ijcard.2014.10.139. Epub 2014 Oct 23. PMID 25464257
- [Background] Gonzalo N, Serruys PW, Okamura T, Shen ZJ, Onuma Y, Garcia-Garcia HM, Sarno G, Schultz C, van Geuns RJ, Ligthart J, Regar E. Optical coherence tomography assessment of the acute effects of stent implantation on the vessel wall: a systematic quantitative approach. Heart. 2009 Dec;95(23):1913-9. doi: 10.1136/hrt.2009.172072. Epub 2009 Aug 10. PMID 19671534
- [Derived] Vilchez-Tschischke JP, Salazar C, Gil-Romero J, Mori R, Nunez-Gil I, Quiros A, Nombela L, Del Trigo M, Jimenez-Quevedo P, Salinas P, Escaned J, Macaya C, Gonzalo N. Stent strut thickness and acute vessel injury during percutaneous coronary interventions: an optical coherence tomography randomized clinical trial. Coron Artery Dis. 2021 Aug 1;32(5):382-390. doi: 10.1097/MCA.0000000000000943. PMID 32826450